CLINICAL TRIAL: NCT01842958
Title: A Randomized, Controlled, Multi-center Clinical Study Evaluating the Crestal Bone Level Changes of Straumann BL Ø 3.3 mm NC SLActive RXD Implants Compared to Straumann BL Ø 4.1 mm RC SLActive RXD Implants for Single Tooth Replacement.
Brief Title: Straumann Roxolid Multi-Center Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR 10/09
Record Dates: First submitted 2013-04-23; First posted 2013-04-30 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-01

CONDITIONS: Jaw, Edentulous, Partially
Keywords: Dental Implant
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4.1 mm implant diameter (Active Comparator): Placement of a Straumann Bone Level Implants, 4.1 mm implant diameter, for single tooth replacement in the anterior and pre-molar region
  Interventions: Device: Straumann Bone Level Implants, 4.1 mm implant diameter
- 3.3 mm implant diameter (Experimental): Placement of a Straumann Bone Level Implants, 3.3 mm implant diameter, for single tooth replacement in the anterior and pre-molar region
  Interventions: Device: Straumann Bone Level Implants, 3.3 mm implant diameter

INTERVENTIONS:
Device: Straumann Bone Level Implants, 4.1 mm implant diameter — Straumann Bone Level Implants, 4.1 mm implant diameter
  Arms: 4.1 mm implant diameter
Device: Straumann Bone Level Implants, 3.3 mm implant diameter — Straumann Bone Level Implants, 3.3 mm implant diameter
  Arms: 3.3 mm implant diameter

SUMMARY:
The primary objective of this study is to demonstrate non-inferiority of the Straumann Bone Level Ø 3.3 mm NC SLActive Roxolid Implants compared to Straumann Bone Level Ø 4.1 mm RC SLActive Roxolid Implants based on mean crestal bone level changes measured between surgery and 12 months post-implant placement. The secondary objectives will assess differences in clinical outcomes between the test and control implants, including implant success and survival, gingival recession, subject satisfaction and additional early bone level measurements.

DETAILED DESCRIPTION:
This is a randomized, controlled, multi-center clinical study. The total study duration for each patient should be 12 ± 1 months.

Straumann Bone Level implants will be placed in the pre-molar or anterior region of the mandible or maxilla for single tooth replacement, followed by provisional prosthetic loading after 25 ± 4 days and by final prosthetic loading 6 ± 1 months after implant loading.

In total 6 visits per patient are scheduled in this study. Bone level changes, implant success and survival, gingival recession, subject satisfaction and adverse events (AEs) will be assessed.

The study devices are CE-(Conformité Européenne, meaning European Conformity) marked products. Straumann Bone Level implants Ø 3.3 mm NC SLActive Roxolid and Straumann Bone Level Ø 4.1 mm RC SLActive implants.

Five centers in USA will participate.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have voluntarily signed the informed consent form
* Subjects must be males or females who are a minimum of 20 years of age
* Subjects must have a single tooth gap in the pre-molar or anterior region of the mandible or maxilla (ADA tooth positions 4-13 and 20-29; FDI tooth positions 11-15, 21-25, 31-35, and 41-45)
* Subjects must have opposing dentition (natural teeth, fixed or removable restorations)
* Subjects must have a full mouth plaque score ≤ 25%, according to O'Leary, at the time of screening
* Subjects must have adequate bone to encapsulate the implant and allow placement of an Ø 4.1 mm Bone Level Implant.
* Adequate bone height of at least 1 mm longer than the length of the study implant
* Subjects must have substantially healed (at least 16 weeks after tooth extraction) extraction sockets
* Subjects must be committed to the study and the required follow-up visits
* Subjects must be in good general health as assessed by the Investigator

Exclusion Criteria:

* Subjects with a systemic disease that would preclude dental implant surgery (e.g. serious internal medical problems, disorders of bone metabolism, uncontrolled bleeding disorders, weakened immune system, illness requiring periodic use of steroids, uncontrollable endocrine disorders, uncontrolled diabetes)
* Subjects with any contraindications for oral surgical procedures (e.g. inadequate wound healing capacity, poor oral hygiene, maxillary and mandibular growth not completed, xerostomia)
* Subjects with mucosal diseases (e.g., erosive lichen planus) in the localized area around the study implant site
* Subjects with a history of local irradiation therapy in the head/neck area
* Subjects with any untreated endodontic lesions or untreated periodontal disease adjacent to the implant site
* Subjects receiving, or having a history of receiving, intravenous or subcutaneous antiresorptive agents, such as bisphosphonates
* Subjects with severe bruxing, parafunctional habits, or temporomandibular joint dysfunction
* Subjects with existing implants in the adjacent positions to the planned implant site
* Subjects requiring bone augmentation or socket grafting within 6 months prior to surgery
* Subjects requiring more than minimal simultaneous augmentation for minimal buccal dehiscence defects (defect cannot be greater than 3mm in height)
* Subjects with inadequate oral hygiene or who are unmotivated for adequate home care
* Subjects who have physical or mental handicaps that would interfere with the ability to perform adequate oral hygiene
* Subjects who are pregnant or intending to become pregnant during the duration of the study
* Subjects who are heavy smokers (defined as >10 cigarettes per day or >1 cigar per day) or chew tobacco
* Subjects who abuse alcohol or drugs
* Subjects who have undergone administration of any investigational device within 30 days of enrollment in the study
* Subjects with conditions or circumstances, in the opinion of the Investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance or unreliability

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-03; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L. Cochran, DDS, MS, PhD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (5):
- United States (5):
  - UCLA School of Dentistry, Los Angeles, California
  - Boston University, School of Dental Medicine, Boston, Massachusetts
  - New York University College of Dentistry, New York, New York
  - Univeristy of Texas Health Science Center San Antonio, San Antonio, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 3.3 mm Implant Diameter: Placement of a Straumann Bone Level Implant, 3.3 mm implant diameter, for single tooth replacement in the anterior and pre-molar region
- 4.1 mm Implant Diameter: Placement of a Straumann Bone Level Implant, 4.1 mm implant diameter, for single tooth replacement in the anterior and pre-molar region
Period: Overall Study
Arm/Group | 3.3 mm Implant Diameter | 4.1 mm Implant Diameter
Started | 25 | 25
Randomized | 25 (One subject was randomized to 3.3 mm implant, but received the 4.1 mm implant.) | 25
Completed | 24 | 24
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population. One subject was randomized to the 3.3 mm implant, but received the 4.1 mm implant. This subject was analyzed according to the actual implant received for the Safety Population/Demographics.
Groups:
- Total: Total of all reporting groups
Arm/Group | 3.3 mm Implant Diameter | 4.1 mm Implant Diameter | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One subject was randomized to the 3.3 mm implant, but received the 4.1 mm implant. This subject was analyzed according to the actual implant received for the Safety Population/Demographics.
  years | 52.9 (13.96) | 49.6 (14.20) | 51.2 (14.04)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject was randomized to the 3.3 mm implant, but received the 4.1 mm implant. This subject was analyzed according to the actual implant received for the Safety Population/Demographics.
  Participants
    Female | 15 | 17 | 32
    Male | 10 | 8 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One subject was randomized to the 3.3 mm implant, but received the 4.1 mm implant. This subject was analyzed according to the actual implant received for the Safety Population/Demographics.
  Participants
    Hispanic or Latino | 3 | 4 | 7
    Not Hispanic or Latino | 22 | 21 | 43
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One subject was randomized to the 3.3 mm implant, but received the 4.1 mm implant. This subject was analyzed according to the actual implant received for the Safety Population/Demographics.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 7 | 5 | 12
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 1 | 2
    White | 16 | 19 | 35
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants] — Population: One subject was randomized to the 3.3 mm implant, but received the 4.1 mm implant. This subject was analyzed according to the actual implant received for the Safety Population/Demographics.
  Participants
    United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Mean Crestal Bone Level Change
Description: Mean crestal bone level change between implant placement and 12 months post loading as determined by radiographic measurement of mesial and distal bone levels following placement of a Straumann Bone Level implant with 3.3 mm diameter versus a Straumann Bone Level implant with 4.1 mm diameter in the anterior or pre-molar region of the mandible or maxilla.
Time Frame: Baseline (implant placement) and 12 months post loading
Population: modified Intent-to-Treat population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 3.3 mm Implant Diameter | 4.1 mm Implant Diameter
Number analyzed (Participants) | 26 | 24
mm | 0.27 (0.34) | 0.48 (0.67)
Statistical Analysis 1: Comparison: 3.3 mm Implant Diameter vs 4.1 mm Implant Diameter; The primary efficacy endpoint is change in crestal bone level from loading to 12 months post-loading. The primary analysis is a test for non-inferiority of the test implant to the control implant at the one-sided 5% significance level. The null hypothesis is that µ3.3 ≥ µ4.1 + δ, where µ3.3 is the mean change in crestal bone level for the test implants, µ4.1 is the mean change in crestal bone level for control implants, and δ is a pre-specified clinically significant difference; Test type: Non-Inferiority — The test arm will be considered non-inferior to the control arm if the 95% upper confidence interval of the estimated difference between the test and control arms is less than -0.5mm; p = 0.02, ANCOVA

2. Secondary Outcome: Additional Mean Crestal Bone Level Changes
Description: Additional radiographic evaluation of mesial and distal crestal bone level changes between implant placement and at 25 days post post implant placement, 6 months post loading, and 12 months post loading
Time Frame: Baseline (implant placement), 25 days post implant placement, 6 months post loading, and 12 months post loading
Population: modified Intent-to-Treat population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 3.3 mm Implant Diameter | 4.1 mm Implant Diameter
Number analyzed (Participants) | 26 | 24
mm
  Change surgery to loading | 0.08 (0.15) | 0.34 (0.38)
  change surgery to 6 months | 0.52 (0.53) | 0.73 (0.52)
  change surgery to 12 months | 0.35 (0.33) | 0.83 (0.66)

3. Secondary Outcome: Implant Success Rate
Description: Percentage of participants with successful and non-successful implant (definition of implant success according to Buser et al. 1991: Absence of persistent subjective complaints, such as pain, foreign body sensation and/ or dysesthesia; Absence of a recurrent peri-implant infection with suppuration; Absence of mobility; Absence of a continuous radiolucency around the implant)
Time Frame: 25 days, 6 months post loading, and 12 months post loading
Population: modified Intent-to-Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | 3.3 mm Implant Diameter | 4.1 mm Implant Diameter
Number analyzed (Participants) | 26 | 24
Participants
  25 days (implant loading): Successful implant | 25 | 23
  25 days (implant loading): Non successful implant | 1 | 1
  25 days (implant loading): Not available for evaluation | 0 | 0
  6 months post loading: Successful implant | 26 | 23
  6 months post loading: Non successful implant | 0 | 0
  6 months post loading: Not available for evaluation | 0 | 1
  12 months post loading: Successful implant | 24 | 24
  12 months post loading: Non successful implant | 0 | 0
  12 months post loading: Not available for evaluation | 2 | 0

4. Secondary Outcome: Implant Survival Rate
Description: Percentage of participants with surviving implant (a surviving implant is one that is in place at the time of follow-up)
Time Frame: 7 days, 25 days, 6 months post loading, and 12 months post loading
Population: modified Intent-to-Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | 3.3 mm Implant Diameter | 4.1 mm Implant Diameter
Number analyzed (Participants) | 26 | 24
Participants
  7 days (post-op): Surviving implant | 26 | 24
  7 days (post-op): Non-surviving implant | 0 | 0
  7 days (post-op): Not available for evaluation | 0 | 0
  25 days (implant loading): Surviving implant | 26 | 24
  25 days (implant loading): Non-surviving implant | 0 | 0
  25 days (implant loading): Not available for evaluation | 0 | 0
  6 months post implant loading: Surviving implant | 26 | 23
  6 months post implant loading: Non-surviving implant | 0 | 0
  6 months post implant loading: Not available for evaluation | 0 | 1
  12 months post implant loading: Surviving implant | 24 | 24
  12 months post implant loading: Non-surviving implant | 0 | 0
  12 months post implant loading: Not available for evaluation | 2 | 0

5. Secondary Outcome: Gingival Recession
Description: Soft tissue measurements include:
  CLI = length of the implant crown from highest point of the soft tissue margin to the incisal edge IPm = distance from the top of the papilla to the incisal edge mesial of the implant crown IPd = distance from the top of the papilla to the incisal edge distal of the implant crown CLTm = length of the crown from highest point of soft tissue margin to the incisal edge of the adjacent mesial tooth CLTd = length of the crown from highest point of soft tissue margin to the incisal edge of the adjacent distal tooth
  Reporting change in soft tissue measurements from 6 months post-loading (final restoration) to 12 months post-loading in millimeters.
Time Frame: 6 months to 12 months post loading
Population: Modified Intent-to-Treat population. Data was not available from 4 subjects in the 3.3 mm arm and 3 subjects in the 4.1 arm
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 3.3 mm Implant Diameter | 4.1 mm Implant Diameter
Number analyzed (Participants) | 22 | 21
mm
  CLI: number analyzed (Participants) | 21 | 21
  CLI | 0.1 (1.04) | 0.2 (2.14)
  IPm | -0.9 (1.4) | -0.9 (1.96)
  IPd | -0.5 (1.54) | -0.9 (1.90)
  CLTm | 0.7 (2.59) | 0.1 (2.76)
  CLTd | 0.8 (1.99) | -0.1 (2.53)

6. Secondary Outcome: Number of Participants With Adverse Events and Adverse Device Effects
Description: Adverse events were checked at each study visit at the following time points: Surgical visit, 7 days (post-op), 25 days (implant loading), 6 months post-loading and 12 months post-loading. The incidence of adverse events during the period of the study is reported here, along with the number of adverse events related to device and procedure (includes "possibly related", "probably related" and "related").
Time Frame: Duration of the study from surgical visit to the 12 months post-loading visit
Population: Safety population. One subject was randomized to the 3.3 mm implant, but received the 4.1 mm implant. This subject was analyzed according to the actual implant received for the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.3 mm Implant Diameter | 4.1 mm Implant Diameter
Number analyzed (Participants) | 25 | 25
Participants
  Subjects without adverse events | 18 | 12
  Subjects with one or more adverse events | 7 | 13
  subjects with adverse events related to device | 1 | 5
  Subjects with adverse events related to procedure | 3 | 5

7. Secondary Outcome: Subject Satisfaction
Description: Subject satisfaction will be assessed utilizing Visual Analogs Scales (VAS) for general satisfaction and pain.
  General satisfaction: ranged from 0 (not satisfied) to 100 (highly satisfied) Pain: ranged from 0 (no pain) to 100 (pain)
Time Frame: 12 months post loading
Population: Modified Intent-to-Treat population. Data was not available for 3 subjects in 3.3 mm implant arm and for 2 subjects in the 4.1 mm implant arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 3.3 mm Implant Diameter | 4.1 mm Implant Diameter
Number analyzed (Participants) | 23 | 22
units on a scale
  General Satisfaction | 97.7 (3.03) | 98.2 (3.54)
  Pain | 6.0 (19.75) | 2.7 (8.05)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from implant surgery to 12 months-post loading, around 13 months total.
Arm/Group | 3.3 mm Implant Diameter | 4.1 mm Implant Diameter
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/25
Other Adverse Events (participants affected / at risk) | 7/25 | 13/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3.3 mm Implant Diameter (N=25) | 4.1 mm Implant Diameter (N=25)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3.3 mm Implant Diameter (N=25) | 4.1 mm Implant Diameter (N=25)
Prosthetic related complication (Surgical and medical procedures) | 5 (9) | 4 (5)
Pain at implant site (Surgical and medical procedures) | 0 (0) | 1 (1)
Implant hit root of adjacent tooth (Surgical and medical procedures) | 0 (0) | 1 (1)
Minimal bone loss around implant (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Implant mobility (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Radiolucency around implant (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Oral ulcer (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain due to bruxism (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tooth caries (General disorders) | 0 (0) | 1 (1)
Adjacent tooth fracutre (General disorders) | 1 (1) | 0 (0)
Vaginal yeast infection (Infections and infestations) | 0 (0) | 1 (1)
Adaptor broke in implant (Product Issues) | 0 (0) | 1 (1)
Burning sensation on labial mucosa (Nervous system disorders) | 0 (0) | 1 (1)
Post op paraesthesia lower left labial mucosa (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days